CLINICAL TRIAL: NCT01948687
Title: The Role of Real Time Elastography in the Noninvasive Assessment of Liver Fibrosis in Chronic Viral Hepatitis
Brief Title: Real Time Elastography in Liver Fibrosis
Acronym: RT-ELASTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy Craiova (Other)
Collaborators: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Principal Investigator, Dan Gheonea, MD, PhD, MSc Specialist in Gastroenterology, University of Medicine and Pharmacy Craiova
Other Study IDs: RT-ELASTO
Record Dates: First submitted 2013-09-03; First posted 2013-09-24 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Cirrhosis; Chronic Liver Disease
Keywords: real time elastography; hepatitis
MeSH Terms: conditions — Fibrosis; Hepatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1. the control group: healthy adult volunteers
- 2. patients with chronic hepatitis: patients with chronic hepatitis B or C (defined by the presence of serum anti hepatitis C antibody or serum hepatitis B surface antigen)
- 3. liver cirrhosis type B or C: patients with liver cirrhosis type B or C

SUMMARY:
AIM To evaluate the role of real time elastography (ARFI and Hitachi elastography) in noninvasive diagnosis of liver fibrosis in patients with chronic hepatitis

DETAILED DESCRIPTION:
INTRODUCTION

Establishing liver fibrosis grade in patients with chronic viral hepatitis is very important for the prognostic assessment and in making the decision to initiate antiviral treatment. Although the liver biopsy remains the gold standard, recent studies focused on establishing the role of noninvasive methods in liver fibrosis grading.

Elastography is an imaging method which estimates tissue elasticity. The first elastography method which appeared was Transient Elastography (TE), followed by Real Time Elastography (RT-E) and Acoustic Radiation Force Impulse (ARFI). TE was a method especially developed for noninvasive assessment of liver fibrosis as an alternative to liver biopsy. Unlike these, RT-E and ARFI have multiple applications in diffuse and tumoral pathology.

Transient Elastography (FibroScan) represents a noninvasive method useful in detecting the degree of liver fibrosis. The ultrasound transducer probe is able to generate elastic shear waves that propagate through the liver tissue as well as to measure their speed in the tissue. Wave speed is directly related to tissue stiffness which is expressed in kilopascals [1]. Initially, this method was validated for use and considered for chronic hepatitis management guidelines, then for human immunodeficiency virus/hepatitis C virus (HCV) co-infection and cholestatic liver diseases. FibroScan failures to give reliable results in obese patients were reduced by developing a new XL probe which facilitated an alternative noninvasive method to liver biopsy for liver fibrosis assessment [2].

Acoustic Radiation Force Impulse (ARFI) was proposed as an alternative to FibroScan for the assessment of liver tissue elasticity, using a conventional ultrasound machine. The main advantages of this method are the possibility of producing real-time images and its feasibility in patients with ascites. Preliminary studies show better results for predicting advanced grades of liver fibrosis than for mild to moderate fibrosis where the method is less sensitive [3].

Real Time Elastography (RT-E) estimates relative tissue stiffness based on soft tissue distortion and data are provided as real time color images [4, 5]. This is a real time method that could also be used for patients with ascites. The method is not validated for liver fibrosis assessment as there are few studies published so far. The appearance of the elastography software on the convex probe with high penetration and possibility for elastography to visualize the liver entirely and the development of information elastography measurement information programs open new perspectives in noninvasive assessment of liver pathology by RT-E. There are two recent studies showing good results of the software for quantitative analysis in RT-E equipment.

The aim of this study is to establish the role of elastographic methods (ARFI and RT-E) in liver fibrosis assessment in patients with chronic viral hepatitis. This multicentric prospective trial will be approved by the ethical committee of each centre.

AIM To evaluate the role of real time elastography (ARFI and Hitachi elastography) in noninvasive diagnosis of liver fibrosis in patients with chronic hepatitis.

MATERIAL AND METHODS

* All patients are enrolled consecutively.
* Patient data are collected (name initials, age, sex, Civil Registration Number), liver disease etiology, anthropometric data (body mass index).
* The following blood parameters are included: aspartate aminotransferase (AST), alanine aminotransferase (ALT), γ -glutamyl transpeptidase, γ globulins, platelet count
* The following indices are calculated: AST/ALT; AST-to-platelet ratio index (APRI); AST/upper limit of normal 100/platelet count (104 /mm3 ) , and FibroIndex [1.738 0.064 x platelet count (104 /mm3 ) + 0.005 x AST (U/l) + 0.463 x γ -globulin (g/dl)]
* Transient elastography is performed using FibroScan (FibroScan, Echosens) with the patient lying in the dorsal decubitus position and with his right arm in maximum abduction. The tip of the transducer probe is placed in the median axillary line in the intercostal space corresponding to the right lobe of the liver. The pressure index on the screen indicates that the pressure applied with the probe is compatible with the measurement. Ten measurements per examination are necessary for good accuracy of the stiffness assessment, considering the final result expressed in kilopascals as the mean of the ten measurements. M and XL probes for obese patients are used.
* Hitachi Real Time Ultrasound Elastography is performed using the 5-1 MHz (EUP) convex transducer from Hitachi Preirus equipment (Hitachi Aloka Medical Tokyo, Japan). Dual imaging is set in such a manner as to be visible on the screen in a 2D image as well as in an elastographic image juxtaposed over the 2D image. The examination is underwent through two points: intercostally through the right lobe and epigastrically through left hepatic lobe. The examination is done through post-expiratory apnea without compression on the probe. The interest region (ROI) is set at 4cm², 1 cm under the liver capsule. The aria of interest is chosen so that the 2D image is as clear as possible, the large vessels avoided and the artifacts given by ribs and lungs. For each patient, 10 images are chosen with two entry points (intercostally and epigastrically). For each image the 11 parameters given by the Strain Histogram measurement software are used: mean relative strain value (MEAN); standard deviation of relative strain value (SD); percentage of low strain area (percentage of blue color area - %AREA); complexity of low strain area (calculated as perimeter 2 /area - COMP); skewness (SKEW); kurtosis (KURT); contrast (CONT); entropy (ENT); textural complexity, inverse difference moment (IDM); angular second moment (ASM); Correlation (CORR) indicates the feature value of the texture directivity.
* ARFI- Acoustic Radiation Force Impulse Technology [ACUSON S2000]. Scanning is performed with a right intercostal approach, in the right liver lobe, segment V-VIII, 1-2 cm under the liver capsule, with minimal scanning pressure applied by the operator, while the patients is asks to stop normal breathing for a moment, in order to minimize breathing motion. The operator selects the depth at which the liver elasticity is evaluated by placing a "measuring box" (10 mm long, 5 mm wide) in the desired area. The maximum depth at which ARFI measurements can be performed is 8 cm. A total of 10 valid measurements performe in every patient and a median value in m/s is calculate.
* Liver biopsy samples is takes via a right intercostal space from the right liver lobe with direct sonographic guidance. Liver fibrosis stages is evaluate semiquantitatively according to the METAVIR scoring system on an F0-F4 scale

Statistical analysis

The diagnostic performance of ARFI and RT-E for liver fibrosis will determine in terms of sensitivity, specificity, positive predictive value, negative predictive value, diagnostic accuracy and area under the receiver operating characteristic curve (AUROC).

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* Study will include three groups of patients as follows:

  1. Group I: patients with chronic hepatitis B or C (defined by the presence of serum anti HCV antibody or serum hepatitis B surface antibody)
  2. Group II (the control group): healthy adult volunteers
  3. Group III: patients with hepatic cirrhosis type B or C
* There at least one reference method available for patients with chronic hepatitis (Transient elastography/ liver biopsy)
* Hepatic cirrhosis diagnosis is established using clinical and paraclinical features (ultrasonography, superior digestive endoscopy)
* A written informed consent is given to each patient

Exclusion Criteria:

* Patients with contraindication for elastography (pregnant women or who are breastfeeding) and patients with pacemakers
* Patients with liver disease of other etiology than viral infection (autoimmune hepatitis, primary biliary hepatitis, primary sclerosing cholangitis, hemochromatosis, alfa 1-antitrypsin deficiency, or Wilson's disease)
* History of alcohol abuse (alcohol intake> 20g/day)
* Patients under treatment with hepatotoxic drugs (methotrexate, amiodarone, corticotherapy , chemotherapy, hormonotherapy)
* Patients with technically unfeasible TE: patients with ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients included in the study will be healthy voluntaries, patients with chronic hepatitis B or C and patients with liver cirrhosis. ARFI and Hitachi elastography will be performed for each patient and the results will be compared with final diagnosis. The final diagnosis (the stage) will be established based on Transient elastography and or liver biopsy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-03 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Real Time Elastography result | up to 24 weeks
  Value of real time elastography recordings for the evaluation of liver fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Saftoiu, MD, PhD, Principal Investigator — UMF Craiova
Locations (2):
- Romania (2):
  - Researche Center of Gastroenterology and Hepatology, Craiova, Dolj
  - University of Medicine and Pharmacy, Timișoara, Timiș County

REFERENCES:
- [Background] 1. Castera L, Forns X, Alberti A. Non-invasive evaluation of liver fibrosis using transient elastography. J Hepatol. 2008; 48: 835-847. 2. V de Lédinghen, Vergniol J, Foucher J, El-Hajbi F, Merrouche W, Rigalleau V. Feasibility of liver transient elastography with FibroScan using a new probe for obese patients. Liver Int. 2010 Aug; 30 (7): 1043-8. 3. Friedrich-Rust M, Nierhoff J, Lupsor M, et al. Performance of Acoustic Radiation Force Impulse imaging for the staging of liver fibrosis: a pooled meta-analysis. J Viral Hepat. 2012 Feb; 19 (2): 212-9. 4. Koizumi Y, Hirooka M, Kisaka Y et al. Liver fibrosis in patients with chronic hepatitis C: noninvasive diagnosis by means of real-time tissue elastography--establishment of the method for measurement. Radiology. 2011; 258: 610-617. 5. Gheonea DI, Săftoiu A, Ciurea T et al. Real-time sono-elastography in the diagnosis of diffuse liver diseases. World J Gastroenterol. 2010; 16: 1720-1726.